CLINICAL TRIAL: NCT07036341
Title: Rehabilitation After a Hip Fracture: the Effects of Dietary Protein and Exercise on Bone and Muscle Health and Quality of Life
Acronym: ProBUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Rijnstate Hospital (Other); Gelderse Vallei Hospital (Other); HAN University of Applied Sciences (Other); Liemerije Revalidatiezorg (Unknown); Opella Revalidatiezorg (Unknown); Pleyade Revalidatiezorg (Unknown); Attent Zorg en Behandeling (Unknown); Alliantie Voeding in de Zorg (Unknown); Osteoporosis Association (Unknown)
Responsible Party: Principal Investigator, Lisette de Groot, prof.dr.ir., Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL68932.081.19
Record Dates: First submitted 2025-05-09; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Hip Fractures
Keywords: Hip fracture patients; Protein; Resistance Exercise; Bone health; Muscle health
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: A randomized controlled two-arm parallel trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group receives a tailor-made protein-enriched diet and an extended progressive resistance training program.
  Interventions: Other: Protein-enriched diet; Other: Progressive resistance exercise
- Control (No Intervention): The control group receives usual care.

INTERVENTIONS:
Other: Protein-enriched diet — A protein intake of 1.5 g/kg bodyweight/day. This will be obtained by consuming protein-rich and protein-enriched foods.
  Arms: Intervention
Other: Progressive resistance exercise — The intervention group will perform resistance training during three non-consecutive days with a minimum of 48 hours between the sessions. Subjects will continue the resistance training after discharge for 2 times a week, also with a minimum of 48 hours between sessions until the study period of 3 months is completed. All sessions will be supervised by physiotherapists.
  Arms: Intervention

SUMMARY:
Hip fractures often lead to functional limitations, loss of independence, weight loss and decreased well-being. Only half of the patients regain their functional level and 24% die within the following year. Financial consequences are significant due to costly surgery and long-term care. Hip fracture incidence is expected to increase sharply due to the ageing population, reducing accessibility to and quality of rehabilitation care. Therefore, optimizing treatment is essential.

Previous protein and exercise studies showed improved muscle and bone health in healthy or frail community-dwelling older adults, but effects in older hip fracture patients are not known. Better rehabilitation may improve bone and muscle health, nutritional status, quality of life, lower costs and lower burden for healthcare.

The overall objective is to investigate the effectiveness, costs and cost-effectiveness of a protein-enriched diet and resistance exercise for 3 months compared to usual care on bone and muscle health, and quality of life in older adults recovering from an acute hip fracture.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age ≥ 65 years
* Acute hip fracture
* Able to give written informed consent
* Mentally competent, as judged by the treating physician
* Admission to a rehabilitation centre that participates in this research

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Allergic, intolerant or hypersensitive to milk/lactose (self-reported)
* Not willing to stop using dietary supplements with exception of calcium and vitamin D
* Pathological fracture or periprosthetic fracture
* Abnormal hepatic or renal laboratory parameters, such as estimated glomerular filtration rate (eGFR) <30 ml/min/1,73 m2 (data from hospital)
* Diagnosis of disorders/diseases where a high protein intake can be harmful, such as renal impairment or failure, or liver disease (geriatric care physician has the decisive voice)
* Diagnosis of bone metabolic disorders such as primary hyperparathyroidism, Paget's disease, or myeloma.
* Taking medication other than bisphosphonates known to strongly alter bone, calcium or muscle metabolism, such as oestrogen, hormone replacement therapy, corticosteroids, anabolic agents, or calcitonin.
* Disorders/diseases which may affect ability to follow study protocol and which cannot be overcome with help of a caregiver
* Current participation in other scientific research
* No permission to request information from the general practitioner/ treating specialist(s) about medical history, medication use, liver and kidney values, and details about the broken hip

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Physical Functioning | Physical performance measurements will be performed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  The short physical performance battery (SPPB) is used to assess physcial functioning. This test is a performance test assessing lower extremity function using measures of gait speed (over 4 meter), standing balance, and lower extremity strength.

SECONDARY OUTCOMES:
Handgrip strength | Handgrip strength will be measured at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  Handgrip strenght will be measured with a hand dynamometer (kg).
Muscle mass | The DEXA scans will be performed at baseline and after 3 months.
  Muscle mass will be quantified using dual-energy X-ray absorptiometry (DEXA).
Bone Mineral Density | The DEXA scans will be performed at baseline and after 3 months.
  BMD will be measured at baseline and after 3 months in the hospital. Total hip, femoral neck and total body BMD (g/cm2) will be measured using DEXA. The unfractured hip will be assessed.
Bone Mineral Density | The quantitative ultrasound measurements will be performed at baseline and after 3 months.
  Quantitative ultrasound (QUS) parameters of the calcaneus will be measured using the portable Achilles EXPII bone ultrasonometer.
Quality of life | Quality of life will be assessed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  Quality of life will be assessed with the EQ5D-5L questionnaire.
Blood markers | Blood markers will be measured at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  Blood markers P1NP, IGF-1, PTH and vitamin D will be measured in serum.
Inpatient rehabilitation time | Assessed at discharge from the rehabilitation centre (varies per participant, on average after 1 month).
  Number of days the patient stayed in the rehabilitation centre.
Daily life functioning | Daily life functioning will be assessed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  The Barthel Index of Activities of Daily Living will be used to assess daily life functioning.
Nutritional Status | This measurement will be performed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  The Mini Nutritional Assessment (MNA) will be used to evaluate nutritional status.
Costs | This will be assessed after 3 months.
  Participants will use a cost diary to keep track of their health care use, out-of-pocket costs, and productivity losses. A health care use questionnaire based on the iMTA Medical Cost Questionnaire will be used, which includes cost categories that were deemed relevant for older adults (general practitioner, home care, informal care, dietitian, physiotherapist, occupational therapist, hospitalization, residential care, rehabilitation care, outpatient clinic, and medication use). Out-of-pocket costs includes sports club memberships, purchase of sport equipment, and other out-of-pocket payments related to the intervention. Productivity losses will be measured using questions from the Productivity Cost Questionnaire.

OTHER OUTCOMES:
Dietary intake | This measurement will be performed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  The dietary intake will be observed and recorded over a period of three non-consecutive days.
Frailty status | This measurement will be performed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  Frailty status is assessed with the Fried criteria.
Body weight | This measurement will be performed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  Body weight in kg
Blood markers | This measurement will be performed at baseline and after 3 months.
  Levels of free vitamin D, folate, vitamin B12 and vitamin C are measured
Physical Activity | This is assessed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  The LASA Physical Activity Questionnaire (LAPAQ) is used to measure physical activity levels.
Appetite | This is assessed at baseline, after discharge from the rehabilitation centre (varies per participant, on average after 1 month), and after 3 months.
  The Simplified Nutritional Appetite Questionnaire (SNAQ) is used to assess appetite.
Fear of falling | This will be assessed after 3 months.
  Fear of falling will be assessed with the Falls Efficacy Scale International (FES-I).
Oral health | This measurement will be performed at baseline.
  Questionnaire
Number of and time to new falls and fragility fractures | This is assessed after 3 months.
  Number of and time to new falls and fragility fractures is assessed with a questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - Gelderse Vallei Hospital, Ede